CLINICAL TRIAL: NCT04777110
Title: The Effectiveness and Safety of Esketamine in Modified Electroconvulsive Therapy for Depressive Patients-- A Multi-center, Randomized , Single-blind Clinical Study
Brief Title: The Effectiveness and Safety of Esketamine in Modified Electroconvulsive Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, Director of Department of Anesthesiology, The First Affiliated Hospital of Chongqing Medical University, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESK-ECT20210222
Record Dates: First submitted 2021-02-22; First posted 2021-03-02 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Esketamine; ECT; Depression
MeSH Terms: conditions — Depression | interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine injection group (0.25mg/kg) (Experimental): The main anesthesiologist standing on the right side of the patient gave successive injections of esketamine (0.25 mg/kg), and 1 minute later, injected propofol (1.5 mg/kg) for 30 s
  Interventions: Drug: Esketamine
- Saline injection group(0.05ml/kg) (Sham Comparator): The main anesthesiologist standing on the right side of the patient sequentially injects normal saline (0.05ml/kg), and 1 minute later injects propofol (1.5 mg/kg), the injection time is 30 seconds
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Esketamine — The main anesthesiologist standing on the right side of the patient injects esketamine (0.25 mg/kg) sequentially, and then propofol (1.5 mg/kg) is injected 1 minute later for 30 s;
  Arms: Esketamine injection group (0.25mg/kg)
Other: Saline — The main anesthesiologist standing on the right side of the patient injects saline (0.05ml/kg) sequentially, and then propofol (1.5 mg/kg) is injected 1 minute later, the injection time is 30 s
  Arms: Saline injection group(0.05ml/kg)

SUMMARY:
A multicenter, randomized, controlled, single blind clinical trial on the efficacy and safety of esmketamine injection in electroconvulsive therapy

Objective to evaluate the efficacy and safety of esmketamine injection in the treatment of non convulsive electroconvulsive therapy

Participants: Patients with depression receiving MECT

The research drug was esketamine injection

The study design was a multicenter, randomized, single blind, parallel controlled trial

25 mg / kg as the experimental group. The normal saline group was the control group (0.05 ml / kg).

The sample size was estimated according to the main efficacy index (remission rate) of this study. It was assumed that the remission rate of the esketamine injection group was better than that of the control group. The parameters were set as test level α = 0.05, unilateral, β = 0.8, the cut-off value was 6%, the experimental group: the control group was 1:1, according to the results of previous clinical trials and combined with literature, the remission rate of the control group was 69%, 159 cases in each group, considering the 20% shedding rate, 198 cases in the experimental group and 198 cases in the control group were selected.

1. experimental group

   The patients were given intravenous injection of 0.25 mg / kg esketamine, 1.5 mg / kg propofol and 1 mg / kg succinylcholine in turn. After anesthesia, the patients were given electroconvulsive therapy
2. In the control group

The patients were given 0.05ml/kg of normal saline, 1.5mg/kg of propofol and 1mg / kg of succinylcholine. After anesthesia, the patients were given electroconvulsive therapy

Efficacy evaluation 1. Main efficacy indicators

Remission rate of depressive symptoms after MECT treatment

Remission was defined as two consecutive hdrs-24 scores ≤ 10 after receiving MECT

Definition rate of remission rate: the proportion of patients with remission of depressive symptoms in this group

ELIGIBILITY:
Inclusion Criteria:

1. Depressed patients receiving MECT for the first time;
2. 16≤age≤45 years old, no gender limit;
3. The ASA score is I or II;
4. Meet the diagnostic criteria for depression established by APA, and the Hamilton Depression Rating Scale (HDRS-24) score ≥ 35 points;
5. The depressive episode lasts at least 2 weeks;
6. Clearly understand and voluntarily participate in the study, and sign an informed consent form.

Exclusion Criteria:

1. Combined with serious physical diseases, such as uncontrolled hypertension, coronary heart disease, intracranial vascular malformations, asthma attacks, severe liver and kidney dysfunction, etc.
2. There are foreign bodies in the body: such as pacemakers, intracranial electrodes, etc.
3. Those with a history of epilepsy
4. Those who are taking reserpine
5. Acute and systemic infectious diseases, moderate or higher fever
6. History of manic episodes
7. Those who are allergic to anesthetics and muscle relaxants
8. Pregnant women
9. Glaucoma
10. Bipolar disorder, or other mental illnesses, mental retardation
11. Those who judged by the physician in charge to be unsuitable for MECT treatment
12. History of drug abuse

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 396 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Relief rate of depressive symptoms after MECT treatment | immediately after the end of each ECT procedure
  After the patient received MECT treatment, the HDRS-24 score ≤ 10 points for two consecutive times

SECONDARY OUTCOMES:
HDRS-24 score after each MECT | Immediately after the end of ECT, four months and six months after the end of the entire treatment course
  HDRS-24 score after each MECT
Treatment response rate | through treatment completion, an average of 18 days
  Response is defined as two consecutive HDRS-24 scores ≤ 50% before treatment after receiving MECT treatment. Effectiveness is defined as the proportion of patients in the group that are treated effectively
Severe suicidal tendency elimination rate | through treatment completion, an average of 18 days
  Severe suicidal tendency is defined as the suicide item score in HDRS-24 ≥ 3 points. The elimination rate of severe suicidal tendency was defined as the proportion of patients with suicide score=0 after treatment in the proportion of patients with severe suicidal tendency
Treatment re-ignition rate | within 4 months of patients in remission
  Re-ignition is defined as an increase in HDRS-24 score of ≥ 10 points within 4 months of patients in remission. The re-ignition rate is defined as the proportion of re-ignition patients in remission patients.
Treatment recurrence rate | up to 4 months
  The HDRS-24 score increased by ≥10 points after 4 months for patients whose recurrence is positioned as remission. The recurrence rate is defined as the proportion of relapsed patients in remission.
Changes in cognitive function | Immediately after the end of ECT, four months and six months after the end of the entire treatment course
  Montreal Cognitive Scale (MoCA) assessment